CLINICAL TRIAL: NCT05887986
Title: Management of Pulmonary Toxicity-related Dyspnea: Effect of Hand-held Fan Airflow Stimulation
Brief Title: Management of Dyspnea: Use of Hand Held Fan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysegul Celik (Other)
Responsible Party: Sponsor-Investigator, Aysegul Celik, Ass. Prof, Izmir Bakircay University
Organization: Izmir Bakircay University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BU
Record Dates: First submitted 2023-04-18; First posted 2023-06-05 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer
Keywords: lung cancer; dyspnea; fan therapy; comfort; oncology nursing
MeSH Terms: conditions — Lung Neoplasms; Dyspnea

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hand-held fan airflow stimulation (Experimental)
  Interventions: Other: hand-held fan airflow stimulation
- control group (No Intervention)

INTERVENTIONS:
Other: hand-held fan airflow stimulation — Outcome dyspnea measures:
  After the fan training application given to the hand-held fan airflow stimulation group by the researchers, the hand fan application will be made for 5 days. On the "baseline", "day 3", and "day 5" of the study, the dyspnea level will be evaluated.
  Outcome comfort measures:
  After the fan training application given to the hand-held fan airflow stimulation group by the researchers, the hand fan application will be made for 5 days. On the "baseline", "day 3", and "day 5" of the study, the comfort level of the patients will be evaluated.
  Arms: hand-held fan airflow stimulation

SUMMARY:
This research is planned as a randomized controlled experimental study to determine the effect of air stimulation to the face with a hand fan in the management of dyspnea in lung cancer patients. The universe of the research was carried out between December 2022 and February 2024, Izmir Provincial Health Directorate, University of Health Sciences, Suat Seren Chest Diseases and Surgery Training and Research Hospital will consist of cancer patients. Individuals who meet the sampling selection criteria from the specified universe will constitute the sample of the research. The sample number of the research was determined as a result of the power analysis made with the G*power program. As a result of the power analysis, based on the t-test in independent groups, the minimum number of samples to be taken was 27 people for a group with 1:1 ratio, 0.80 power, effect value 0.80 and 0.05 significance level. Randomization of the sample will be ensured by accepting the first patient who applied to the outpatient chemotherapy unit randomly and with an appointment at the beginning of the study to the experimental group, and the next patient to the control group. Considering the losses, it is planned to work with 60 people, 30 people in the intervention group and 30 people in the control group. Individual Descriptive Information Form, Medical Research Council Scale (mMRC), Cancer Dyspnea Scale, Vital Signs Follow-up Form, Eastern Cooperative Oncology Group (ECOG) Performance Scale and General Comfort Scale Short Form will be used.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Diagnosed with lung cancer
* mMRC dyspnea scale score ≥2
* ECOG Performance Score score ≥3
* Volunteered to participate in the research

Exclusion Criteria:

* Having a fever of 38⁰C and above in the last 24 hours
* Inability to communicate cognitively and verbally
* Having a psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
dyspnea level | baseline, day 3, and day 5
  Cancer Dyspnea Scale: It will be used to evaluate dyspnea level of cancer patient. The scale was developed by Tanaka et al (2000); An adaptation study for Turkish society was made by Bitek and Tokem (2021). The scale consists of 12 items and three dimensions (effort, anxiety, feelings of discomfort). Cronbach's alpha coefficients varying between 0.81 and 0.93 were reported for all three sub-dimensions. Three sub-dimensions and total score values are used in the evaluation of the scale. The scale is scored likert type and 1: None; 2: a little; 3: Quite; 4: Significantly; 5: Shows Too Many expressions. The total score obtained from the scale is 48. The increase in the total score obtained from the scale indicates the increase in the severity of dyspnea.

SECONDARY OUTCOMES:
comfort level | baseline, day 3, and day 5
  General Comfort Scale- Short Form: It was developed by Kolcaba in 2006. The validity and reliability study in our country was carried out by Sarıtaş et al (2018). The scale includes the sub-dimensions of comfort, relief (1-9 items), relaxation (9-18 items) and overcoming problems (1-28 items) from 28 items. These items are evaluated as Likert type ranging from "strongly disagree (1) to "strongly agree (6)". The average value is found by dividing the total score obtained by the number of scale items. The lowest value that can be taken is 1, which indicates a low level of comfort, and the highest value of 6 indicates a high level of comfort. The Cronbach alpha value of the scale was found to be 0.82

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Provincial Health Directorate Health Sciences University Dr. Suat Seren Chest Diseases and Surgery Training and Research Hospital, Izmir, Turkey (Türkiye)